CLINICAL TRIAL: NCT02021513
Title: Pilot Study - Effect of Omega-3 on Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Cristina Gale Arriens, Postdoctural Fellow Clinical Research, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EO3SLE
Record Dates: First submitted 2013-12-13; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Fish Oil; Omega-3
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Fish Oils; Fatty Acids, Omega-3; Olive Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish Oil (Experimental): Fish Oil (2.25gm EPA and 2.25gm DHA total)
  Interventions: Dietary Supplement: Fish Oil
- Placebo (Placebo Comparator): Olive Oil
  Interventions: Dietary Supplement: Olive Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — Fish Oil (2.25gm EPA and 2.25gm DHA total)
  Other Names: Omega-3 Fatty Acids; DHA/EPA
  Arms: Fish Oil
Dietary Supplement: Olive Oil — Placebo group
  Arms: Placebo

SUMMARY:
This is a single blind placebo-controlled pilot study involving Systemic Lupus Erythematosus and lupus nephritis patients. We propose to recruit and consent SLE patients who will be randomized to either receive the study drug, an over the counter fish oil supplement, or a placebo that contains olive oil. They will have a baseline metabolomic profile (blood test), nutritional assessment, fatigue severity scale, quality of life assessment, and SELENA-SLEDAI lupus disease activity assessments completed at the time of study medication distribution. Once 6 months of either the study drug or placebo is completed, then pill counts, assessments of experience/adherence (including side-effects, adverse effects, complaints, and un-blinding), and repeat nutritional assessment, fatigue severity scale, SELENA-SLEDAI, and metabolomic profile will be assessed. The study duration for each patient will be 6 months from initiation of the study drug. It is hypothesized that patients receiving the fish oil supplement will have improvement in their metabolomic profile. Additionally it is hypothesized that patients receiving the fish oil supplement will have improvement in disease activity, fatigue, and quality of life assessments.

DETAILED DESCRIPTION:
Supplementation with EPA and DHA could potentially reduce the inflammatory state of SLE patients. This study is a single blind placebo-controlled pilot for SLE patients with 25 scheduled to receive omega-3 (EPA 2.25g/DHA 2.25g) daily and 25 scheduled to receive placebo (olive oil), for 6 months. Pre and post supplementation assessments will be made to determine if EPA and DHA levels increase, and if the levels of lipid peroxidation products, other cellular energy intermediates, and inflammatory markers are affected by EPA/DHA. Additionally, lupus disease activity, fatigue, quality of life, and diet will be assessed to determine if these parameters are related to the metabolome in SLE.

* Aim 1:

  - To determine if the metabolomic disturbances of lupus patients improve following supplementation with omega-3 fatty acids.
* Aim 2:

  * To determine if lupus disease activity, fatigue, and quality of life improve and are related to the metabolomic profile changes.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* All ethnic groups
* Aged 18-64
* Biopsy proven diagnosis of Lupus Nephritis and/or fulfillment of 4 or more American College of Rheumatology criteria for the diagnosis of Systemic Lupus Erythematosus

Exclusion Criteria:

* Currently taking, or have taken in the last 2 months, fish oil/omega-3 fatty acid/DHA/EPA
* Allergic to fish oil, shellfish, or other fish products
* Pregnant
* Currently taking the medication: Tositumomab (Bexxar)
* Currently taking anti-coagulant medications (Abciximab, Acenocoumarol, Anisindione, Ardeparin, Argatroban, Bivalirudin, Certoparin, Cilostazol, Clopidogrel, Dalteparin, Danaparoid, Defibrotide, Dermatan Sulfate, Desirudin, Dicumarol, Enoxaparin, Eptifibatide, Fondaparinux, Heparin, Lamifiban, Nadroparin, Phenindione, Phenprocoumon, Reviparin, Sibrafiban, Tinzaparin,Tirofiban, Warfarin, Xemilofiban)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Metabolomic profile | Change from baseline at 6 months
  Blood collection by venipuncture for serum assessment of metabolomic profile (fatty acids, markers of oxidative stress, markers of inflammation, markers of energy stores).

SECONDARY OUTCOMES:
Disease Activity | Change from baseline at 6 months
  SELENA-SLEDAI
SF-36 | Change from baseline at 6 months
  RAND Short Form 36 Quality of Life Assessment
FSS | Change from baseline at 6 months
  Fatigue Severity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Cristina G Arriens, MD, Study Chair — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Arriens C, Hynan LS, Lerman RH, Karp DR, Mohan C. Placebo-controlled randomized clinical trial of fish oil's impact on fatigue, quality of life, and disease activity in Systemic Lupus Erythematosus. Nutr J. 2015 Aug 18;14:82. doi: 10.1186/s12937-015-0068-2. PMID 26283629